CLINICAL TRIAL: NCT02207257
Title: Phase II Randomized, Sequential Group, Evaluation of Ascending Reversal Doses of PER977 Administered to Subjects With Steady State Edoxaban Dosing and Re-anticoagulation With Edoxaban Following PER977 Reversal
Brief Title: Study of PER977 Administered to Subjects With Steady State Edoxaban Dosing and Re-anticoagulation With Edoxaban
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Perosphere Pharmaceuticals Inc, a wholly owned subsidiary of AMAG Pharmaceuticals, Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: AMAG Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: PER977-02-001
Record Dates: First submitted 2014-07-28; First posted 2014-08-04 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2017-11

CONDITIONS: Anticoagulation Reversal
Keywords: PER977; anticoagulation reversal; pharmacokinetics; edoxaban; whole blood clotting time; D-dimer; prothrombin fragments 1 and 2; tissue factor pathway inhibitor; prothrombin time
MeSH Terms: interventions — PER977; edoxaban

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 (Experimental): Subjects will receive 60 mg edoxaban in the morning on Days 1-2. On Day 3 and 4, they will receive a single dose of 60 mg edoxaban, followed 3 hours later by a single dose of 25 mg PER977 or placebo (n=10).
  Interventions: Drug: PER977; Drug: Placebo; Drug: Edoxaban
- Cohort 2 (Experimental): Subjects will receive 60 mg edoxaban in the morning on Days 1-2. On Day 3 and 4, they will receive a single dose of 60 mg edoxaban, followed 3 hours later by a single dose of 50 mg PER977 or placebo (n=10).
  Interventions: Drug: PER977; Drug: Placebo; Drug: Edoxaban
- Cohort 3 (Experimental): Subjects will receive 60 mg edoxaban in the morning on Days 1-2. On Day 3 and 4, they will receive a single dose of 60 mg edoxaban, followed 3 hours later by a single dose of 100 mg PER977 or placebo (n=10).
  Interventions: Drug: PER977; Drug: Placebo; Drug: Edoxaban
- Cohort 4 (Experimental): Subjects will receive 60 mg edoxaban in the morning on Days 1-2. On Day 3 and 4, they will receive a single dose of 60 mg edoxaban, followed 3 hours later by a single dose of 300 mg PER977 or placebo (n=10). Study amendments expanded the cohort to include an additional 7 subjects (randomized 1:6 PER977:placebo) and up to an additional 4 placebo and 8 active subjects (ongoing).
  Interventions: Drug: PER977; Drug: Placebo; Drug: Edoxaban
- Cohort 5 (Experimental): Subjects will receive 60 mg edoxaban in the morning on Days 1-2. On Day 3 and 4, they will receive a single dose of 60 mg edoxaban, followed 3 hours later by a single dose of 600 mg PER977 or placebo (n=10). A protocol amendment expanded the cohort to include an additional 2 placebo and up to an additional 4 active subject.
  Interventions: Drug: PER977; Drug: Placebo; Drug: Edoxaban

INTERVENTIONS:
Drug: PER977 — Reversal of edoxaban-induced anticoagulation
Drug: Placebo — Reversal of edoxaban-induced anticoagulation
Drug: Edoxaban

SUMMARY:
This study will evaluate the establishment of anticoagulation ("re-anticoagulation") of subjects with edoxaban following reversal by PER977 and will identify a dose regimen of PER977 that reverses the effects of edoxaban for up to 21 hours.

DETAILED DESCRIPTION:
This is a randomized, single-blind, sequential group, ascending PER977 reversal dose study in healthy volunteers. Subjects will be randomized in a 4:1 ratio to receive either PER977 or placebo. All subjects will receive a single dose of edoxaban 60 mg on Days 1-4. On Days 3 and 4, study drug will be administered 3 hours following edoxaban. Beginning with Cohort 2, study drug will be administered only to those subjects with a minimum increase in whole blood clotting time >25% above baseline.

Pharmacokinetic assessment of PER977 and tis metabolite, and edoxaban and its metabolite will be performed. Pharmacodynamic assessment of WBCT and Point of Care prothrombin time will be performed. Safety will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 to 65 years, inclusive
2. Laboratory values are not clinically significant
3. No clinically significant findings on 12-lead electrocardiogram
4. Body mass index (BMI) 18 to ≤ 32 kg/m2, inclusive
5. Male subjects agree to use appropriate contraception .
6. Female subjects may be post-menopausal or, if of child-bearing potential, must have a negative serum pregnancy test prior to enrollment, and must agree to use two forms of acceptable contraception for the duration of the study and for a minimum of one complete menstrual cycle or 28 days following discharge from the study.
7. Subjects must sign informed consent

Exclusion Criteria:

1. History or current evidence of clinically significant disease, liver function tests greater than the upper limit of normal (presence of Gilbert's syndrome is acceptable), QTcF > normal (440±10 msec for males or 460±10 msec for females).
2. History of unexplained syncope
3. History of major bleeding, trauma, surgical procedure of any type, or vaginal delivery within six months prior to screening
4. History of peptic ulcer, gastrointestinal bleeding, including the mouth, within six months prior to screening
5. History of minor bleeding episodes such as epistaxis, rectal or hemorrhoidal bleeding or gingival bleeding within 1 month prior to screening
6. Personal or family history of clotting disorder or abnormality, excessive bleeding, thrombovascular disease or any hematologic disorder involving platelets or clotting abnormalities or any condition requiring treatment with transfusions, or history of heparin-induced thrombocytopenia
7. Females with a history of dysfunctional uterine bleeding, menorrhagia , metrorrhagia or polymenorrhea
8. Pregnant or breast-feeding
9. Males with a history of hormone therapy within 3 months prior to screening
10. Administration of any blood product or anticoagulant within 3 months prior to study entry or any non steroidal anti-inflammatory drug or cyclooxygenase inhibitor within 2 weeks prior to screening
11. Taking any type of chronic medication within the 4 weeks prior to study entry (use of hormonal contraceptives is acceptable)
12. Positive serologic test for HIV, HCV-Ab, or HBsAG
13. Donation of blood or blood products within 56 days prior to screening
14. Smokers or use of tobacco and/or nicotine containing products within 3 months prior to dosing as determined by the subject's verbal history
15. Participation in any study with an investigational compound or device within 30 days prior to signing informed consent
16. History of participation in any prior study of PER977 or edoxaban
17. Active drug or alcohol dependence within the prior 12 months or any condition that, in the opinion of the Investigator, would interfere with adherence to study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-03; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Whole blood clotting time as a measure of edoxaban anticoagulation reversal by PER977 | 5 days
  To evaluate the safety, tolerability and effect on whole blood clotting time of escalating intravenous doses of PER977 (25, 50, 100, 300 mg, and 600 mg) administered after 60 mg edoxaban as a "rescue" medication in healthy volunteers and repeated for a second day to investigate any effects of PER977 on the re-anticoagulation with edoxaban and second reversal with PER977.

SECONDARY OUTCOMES:
Pharmacokinetic profile of PER977 | 5 days
  To assess the maximal concentration, half-life and plasma and urinary clearance of PER977 and its metabolite following intravenous administration
Pharmacokinetic profile of edoxaban | 5 days
  To evaluate the maximal concentration, half-life, and clearance of edoxaban and its metabolite when administered with PER977
Safety coagulation measures | 5 days
  To evaluate changes in point of care prothrombin time, d-dimer, prothrombin factors 1 and 2, tissue factor pathway inhibitor, and possibly other biomarkers following escalating intravenous doses of PER977 administered after edoxaban in healthy volunteers
Safety and tolerability | 5 days
  To determine if adverse events occurred in healthy volunteers who received PER977 after edoxaban

OTHER OUTCOMES:
Analytical measurement range (AMR), reproducibility, and precision of WBCT measurements | 5 days
  To determine to normal range, variability, and reproducibility of WBCT in blood collected from healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rasmussen, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Quintiles, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Sciascia S, Lopez-Pedrera C, Cecchi I, Pecoraro C, Roccatello D, Cuadrado MJ. Non-vitamin K antagonist oral anticoagulants and antiphospholipid syndrome. Rheumatology (Oxford). 2016 Oct;55(10):1726-35. doi: 10.1093/rheumatology/kev445. Epub 2016 Feb 3. PMID 26843482